CLINICAL TRIAL: NCT01172639
Title: A 2 Year Prospective Multicentre Randomised Controlled Trial Comparing Effectiveness in Daily Practice of Different Treatment Strategies for Early Rheumatoid Arthritis.
Brief Title: Effectiveness in Daily Practice of Different Treatment Strategies for Early Rheumatoid Arthritis.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: P. Verschueren (Other)
Collaborators: Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Sponsor-Investigator, P. Verschueren, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CareRA; 2008-007225-39 (EudraCT Number)
Record Dates: First submitted 2010-07-28; First posted 2010-07-30 (Estimated); Results first posted 2018-12-10 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Rheumatoid Arthritis
Keywords: CoBRA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Sulfasalazine; Salazopyrine; Leflunomide; Prednisone

STUDY DESIGN:
Intervention Model Description: Before randomisation patients were stratified to a high-risk or low-risk group according to the presence of risk factors at screening (having erosions, rheumatoid factor and/or anticitrullinated protein antibody and a high disease activity score calculated with C-reactive protein (DAS28-CRP)). Randomisation to treatment arms was performed via a digitally generated sequence. Patients in the high-risk group were randomised into CoBRA Classic, Clim or Avant-Garde arm. Patients in the low-risk group were randomised into CoBRA Slim or Tight Step Up arm.
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- CoBRA classic high risk group (Other): * Methotrexate 15mg tablet by mouth, weekly for entire trial
  * Sulfasalazine 2g tablet by mouth, daily for 40 weeks
  * Prednisone tablet by mouth, weekly step down scheme 60 - 40 - 25 - 20 - 15 - 10 mg daily for 6 weeks, followed by 7.5mg daily till week 28, then further tapered down to stop at week 32
  Interventions: Drug: Methotrexate; Drug: Sulfasalazine; Drug: Prednisone
- CoBRA slim high risk group (Other): * Methotrexate 15mg tablet by mouth, weekly for entire trial
  * Prednisone tablet by mouth, weekly step down scheme 30 - 20 - 12.5 - 10 - 7.5 mg daily for 5 weeks, followed by 5mg daily till week 28, then further tapered down to stop at week 32
  Interventions: Drug: Methotrexate; Drug: Prednisone
- CoBRA avant-garde high risk group (Other): * Methotrexate 15mg tablet by mouth, weekly for 40 weeks (continued for entire trial if randomized to Methotrexate monotherapy at week 40)
  * Leflunomide 10mg tablet by mouth, daily for 40 weeks (continued for entire trial if randomized to Leflunomide monotherapy at week 40)
  * Prednisone tablet by mouth, weekly step down scheme 30 - 20 - 12.5 - 10 - 7.5 mg daily for 5 weeks, followed by 5mg daily till week 28, then further tapered down to stop at week 32
  Interventions: Drug: Methotrexate; Drug: Leflunomide; Drug: Prednisone
- CoBRA slim low risk group (Other): * Methotrexate 15mg tablet by mouth, weekly for entire trial
  * Prednisone tablet by mouth, weekly step down scheme 30 - 20 - 12.5 - 10 - 7.5 mg daily for 5 weeks, followed by 5mg daily till week 28, then further tapered down to stop at week 32
  Interventions: Drug: Methotrexate; Drug: Prednisone
- Tight Step Up low risk group (Other): * Methotrexate 15mg tablet by mouth, weekly for entire trial
  * No oral steroids allowed during the first year of the trial
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — Methotrexate tablet
  Other Names: Ledertrexate
Drug: Sulfasalazine — Sulfasalazine tablet
  Other Names: Salazopyrine
  Arms: CoBRA classic high risk group
Drug: Leflunomide — Leflunomide tablet
  Other Names: Arava
  Arms: CoBRA avant-garde high risk group
Drug: Prednisone — Prednisone tablet
  Arms: CoBRA avant-garde high risk group; CoBRA classic high risk group; CoBRA slim high risk group; CoBRA slim low risk group

SUMMARY:
The Combinatietherapie Bij Reumatoide Artritis (CoBRA) trial was a milestone in the development of the present treatment paradigm for Rheumatoid Arthritis (RA). This study introduced the principle of fast remission induction by means of a combination of standard Disease Modifying AntiRheumatic Drugs (DMARDs) and a step down bridge therapy with high dose glucocorticoids in early Rheumatoid Arthritis.

The purpose of the present study is to compare different combinations of traditional DMARDs and glucocorticoids, based on the original CoBRA protocol, for treatment of early Rheumatoid Arthritis.

Besides the efficacy and effectiveness of these strategies, patient centered outcomes and potential implementation problems of such treatment strategies are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA as defined by the 1987 or 2010 revised American College of Rheumatology (ACR) criteria
* Early RA (less than 1 year)
* Use a reliable method of contraception for women of childbearing potential
* Able and willing to give written informed consent and participate in the study

Exclusion Criteria:

* Previous treatment with DMARDs
* Previous treatment with oral corticosteroids at a dosage of more than 10 milligrams (mg) prednisone within 4 weeks before baseline
* Previous treatment with oral corticosteroids at a dosage equal to or less than 10 mg prednisone within 2 weeks before baseline
* Previous treatment with oral corticosteroids for more than 4 weeks
* Previous treatment with Intra Articular corticosteroids within 4 weeks before baseline
* Previous treatment with an investigational drug for the treatment or prevention of RA
* Contraindications for corticosteroids
* Contraindications for DMARDs
* Psoriatic Arthritis
* Underlying cardiac, pulmonary, metabolic, renal or gastrointestinal conditions, chronic or latent infectious diseases or immune deficiency which in the opinion of the investigator places the patient at an unacceptable risk for participation in the study
* Pregnancy, breastfeeding or no use of a reliable method of contraception
* Alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2009-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Verschueren, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (17):
- Belgium (17):
  - ASZ, Aalst
  - OLV Ziekenhuis, Aalst
  - Imelda Ziekenhuis, Bonheiden
  - AZ St Lucas, Bruges
  - Reuma praktijk, Genk
  - Reumacentrum, Genk
  - UZ Gent, dept. of Rheumatology, Ghent
  - Reuma instituut Hasselt, Hasselt
  - Reumapraktijk, Hasselt
  - Jan Yperman Ziekenhuis, Ieper
  - AZ groeninge, Kortrijk
  - HHart Ziekenhuis, Leuven
  - MCH, Leuven
  - Universitaire Ziekenhuizen Leuven, Leuven
  - AZ St maarten, Mechelen
  - ZNA Jan Palfijn, Merksem
  - Henri Serruys ziekenhuis, Ostend

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Verschueren P, Esselens G, Westhovens R. Predictors of remission, normalized physical function, and changes in the working situation during follow-up of patients with early rheumatoid arthritis: an observational study. Scand J Rheumatol. 2009 May-Jun;38(3):166-72. doi: 10.1080/03009740802484846. PMID 19169906
- [Background] Verschueren P, Esselens G, Westhovens R. Daily practice effectiveness of a step-down treatment in comparison with a tight step-up for early rheumatoid arthritis. Rheumatology (Oxford). 2008 Jan;47(1):59-64. doi: 10.1093/rheumatology/kem288. Epub 2007 Nov 26. PMID 18039681
- [Background] Durez P, Malghem J, Nzeusseu Toukap A, Depresseux G, Lauwerys BR, Westhovens R, Luyten FP, Corluy L, Houssiau FA, Verschueren P. Treatment of early rheumatoid arthritis: a randomized magnetic resonance imaging study comparing the effects of methotrexate alone, methotrexate in combination with infliximab, and methotrexate in combination with intravenous pulse methylprednisolone. Arthritis Rheum. 2007 Dec;56(12):3919-27. doi: 10.1002/art.23055. PMID 18050189
- [Background] Esselens G, Westhovens R, Verschueren P. Effectiveness of an integrated outpatient care programme compared with present-day standard care in early rheumatoid arthritis. Musculoskeletal Care. 2009 Mar;7(1):1-16. doi: 10.1002/msc.136. PMID 18618520
- [Background] Boers M, Verhoeven AC, Markusse HM, van de Laar MA, Westhovens R, van Denderen JC, van Zeben D, Dijkmans BA, Peeters AJ, Jacobs P, van den Brink HR, Schouten HJ, van der Heijde DM, Boonen A, van der Linden S. Randomised comparison of combined step-down prednisolone, methotrexate and sulphasalazine with sulphasalazine alone in early rheumatoid arthritis. Lancet. 1997 Aug 2;350(9074):309-18. doi: 10.1016/S0140-6736(97)01300-7. PMID 9251634
- [Background] De Cock D, Van der Elst K, Meyfroidt S, Verschueren P, Westhovens R. The optimal combination therapy for the treatment of early rheumatoid arthritis. Expert Opin Pharmacother. 2015;16(11):1615-25. doi: 10.1517/14656566.2015.1056735. Epub 2015 Jun 10. PMID 26058860
- [Result] Verschueren P, De Cock D, Corluy L, Joos R, Langenaken C, Taelman V, Raeman F, Ravelingien I, Vandevyvere K, Lenaerts J, Geens E, Geusens P, Vanhoof J, Durnez A, Remans J, Vander Cruyssen B, Van Essche E, Sileghem A, De Brabanter G, Joly J, Meyfroidt S, Van der Elst K, Westhovens R. Methotrexate in combination with other DMARDs is not superior to methotrexate alone for remission induction with moderate-to-high-dose glucocorticoid bridging in early rheumatoid arthritis after 16 weeks of treatment: the CareRA trial. Ann Rheum Dis. 2015 Jan;74(1):27-34. doi: 10.1136/annrheumdis-2014-205489. Epub 2014 Oct 30. PMID 25359382
- [Result] Verschueren P, De Cock D, Corluy L, Joos R, Langenaken C, Taelman V, Raeman F, Ravelingien I, Vandevyvere K, Lenaerts J, Geens E, Geusens P, Vanhoof J, Durnez A, Remans J, Vander Cruyssen B, Van Essche E, Sileghem A, De Brabanter G, Joly J, Van der Elst K, Meyfroidt S, Westhovens R; CareRA study group. Patients lacking classical poor prognostic markers might also benefit from a step-down glucocorticoid bridging scheme in early rheumatoid arthritis: week 16 results from the randomized multicenter CareRA trial. Arthritis Res Ther. 2015 Apr 9;17(1):97. doi: 10.1186/s13075-015-0611-8. PMID 25889222
- [Result] Verschueren P, De Cock D, Corluy L, Joos R, Langenaken C, Taelman V, Raeman F, Ravelingien I, Vandevyvere K, Lenaerts J, Geens E, Geusens P, Vanhoof J, Durnez A, Remans J, Vander Cruyssen B, Van Essche E, Sileghem A, De Brabanter G, Joly J, Meyfroidt S, Van der Elst K, Westhovens R. Effectiveness of methotrexate with step-down glucocorticoid remission induction (COBRA Slim) versus other intensive treatment strategies for early rheumatoid arthritis in a treat-to-target approach: 1-year results of CareRA, a randomised pragmatic open-label superiority trial. Ann Rheum Dis. 2017 Mar;76(3):511-520. doi: 10.1136/annrheumdis-2016-209212. Epub 2016 Jul 18. PMID 27432356
- [Derived] Pazmino S, Boonen A, De Cock D, Stouten V, Joly J, Bertrand D, Westhovens R, Verschueren P. Short-term glucocorticoids reduce risk of chronic NSAID and analgesic use in early methotrexate-treated rheumatoid arthritis patients with favourable prognosis: subanalysis of the CareRA randomised controlled trial. RMD Open. 2021 May;7(2):e001615. doi: 10.1136/rmdopen-2021-001615. PMID 34031262
- [Derived] Stouten V, Westhovens R, De Cock D, Van der Elst K, Pazmino S, Bertrand D, Joly J, Verschueren P. Having a co-morbidity predicts worse outcome in early rheumatoid arthritis despite intensive treatment: a post hoc evaluation of the pragmatic randomized controlled CareRA trial. Rheumatology (Oxford). 2021 Aug 2;60(8):3699-3708. doi: 10.1093/rheumatology/keaa841. PMID 33434277
- [Derived] Pazmino S, Lovik A, Boonen A, De Cock D, Stouten V, Joly J, Bertrand D, Van der Elst K, Westhovens R, Verschueren P. Does Including Pain, Fatigue, and Physical Function When Assessing Patients with Early Rheumatoid Arthritis Provide a Comprehensive Picture of Disease Burden? J Rheumatol. 2021 Feb;48(2):174-178. doi: 10.3899/jrheum.200758. Epub 2020 Nov 15. PMID 33191282
- [Derived] Pazmino S, Boonen A, Stouten V, De Cock D, Joly J, Van der Elst K, Westhovens R, Verschueren P. Two-year cost-effectiveness of different COBRA-like intensive remission induction schemes in early rheumatoid arthritis: a piggyback study on the pragmatic randomised controlled CareRA trial. Ann Rheum Dis. 2020 May;79(5):556-565. doi: 10.1136/annrheumdis-2019-216874. Epub 2020 Apr 2. PMID 32241795
- [Derived] Stouten V, Michiels S, Westhovens R, De Cock D, Belba A, Pazmino S, Van der Elst K, Joly J, Verschueren P. Effectiveness of maintenance therapy with methotrexate compared with leflunomide for patients with RA having achieved disease control with both these drugs: results of a predefined sub-analysis of CareRA, a pragmatic RCT. Clin Rheumatol. 2020 Sep;39(9):2593-2601. doi: 10.1007/s10067-020-05008-4. Epub 2020 Mar 12. PMID 32166429
- [Derived] Stouten V, Westhovens R, Pazmino S, De Cock D, Van der Elst K, Joly J, Verschueren P; CareRA study group. Effectiveness of different combinations of DMARDs and glucocorticoid bridging in early rheumatoid arthritis: two-year results of CareRA. Rheumatology (Oxford). 2019 Dec 1;58(12):2284-2294. doi: 10.1093/rheumatology/kez213. PMID 31236568

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 400 participants between January 2009 and May 2013. There were 13 participating Flemish rheumatology centers (2 academic centers, 7 general hospitals and 4 private practices).
Pre-assignment Details: There were 379 patients randomised to a treatment arm, 21 patients not randomised: 1 screen failure, 10 withdrawals by subject, 10 randomisation errors
Period: Overall Study
Arm/Group | CoBRA Classic High Risk Group | CoBRA Slim High Risk Group | CoBRA Avant-garde High Risk Group | CoBRA Slim Low Risk Group | Tight Step Up Low Risk Group
Started | 98 | 98 | 93 | 43 | 47
Week 16 | 94 | 96 | 91 | 39 | 47
Week 52 | 89 | 89 | 88 | 38 | 45
Completed | 85 | 87 | 77 | 32 | 41
Not Completed | 13 | 11 | 16 | 11 | 6
Not completed — Death | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 9 | 7 | 11 | 6 | 6
Not completed — Withdrawal by Subject | 3 | 3 | 5 | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- CoBRA Classic High Risk Group: * Methotrexate (MTX)
  * Sulphasalazine
  * Step down steroid full dose
  randomisation: Stratification according to risk factors into two groups. Random assignment to different treatment strategies within strata.
- CoBRA Slim High Risk Group; CoBRA Slim Low Risk Group: * MTX
  * Step down steroid half dose
  randomisation: Stratification according to risk factors into two groups. Random assignment to different treatment strategies within strata.
- CoBRA Avant-garde High Risk Group: * MTX
  * Leflunomide
  * Step down steroid half dose
  randomisation: Stratification according to risk factors into two groups. Random assignment to different treatment strategies within strata.
- Tight Step Up Low Risk Group: * MTX
  * No additional oral steroids allowed
  randomisation: Stratification according to risk factors into two groups. Random assignment to different treatment strategies within strata.
- Total: Total of all reporting groups
Arm/Group | CoBRA Classic High Risk Group | CoBRA Slim High Risk Group | CoBRA Avant-garde High Risk Group | CoBRA Slim Low Risk Group | Tight Step Up Low Risk Group | Total
Number analyzed (Participants) | 98 | 98 | 93 | 43 | 47 | 379
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (11.9) | 51.8 (13.1) | 51.1 (12.8) | 51.4 (14.4) | 51.0 (14.0) | 51.9 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 63 | 64 | 33 | 38 | 262
  Male | 34 | 35 | 29 | 10 | 9 | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 95 | 96 | 90 | 43 | 47 | 371
  Hispanic | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 0 | 0 | 3
  Black | 1 | 1 | 1 | 0 | 0 | 3
  North African | 0 | 0 | 2 | 0 | 0 | 2
Smoking status [Count of Participants; unit: Participants]
  current | 30 | 30 | 23 | 10 | 4 | 97
  past | 26 | 28 | 33 | 11 | 14 | 112
  never | 42 | 40 | 37 | 22 | 29 | 170
Symptom duration [Mean (Standard Deviation); unit: weeks] | 33.8 (35.5) | 33.2 (38.2) | 44.3 (65.9) | 34.4 (68.2) | 33.1 (62.2) | 36.2 (52.6)

OUTCOME MEASURES:

1. Primary Outcome: Remission According to DAS28-CRP at Week 16
Description: Number of patients in remission according to DAS28-CRP (Disease Activity Score based on 28 joint count and C-reactive Protein) at week 16.
  DAS28-CRP is calculated with the following formula : 0.56*SQRT TJC28+0.28*SQRT SJC28+0.36*ln (CRP+1)+0.014*GH+0.96 in which TJC is the tender joint count, SJC the Swollen Joint Count and GH the general health estimated by the patient on a Visual Analogue Scale (VAS).
  A value below 2.6 is indicating remission, below or equal to 3.2 low disease activity, between 3.2 and 5.1 moderate disease activity and above 5.1 high disease activity.
Time Frame: week 16
Population: ITT = intention to treat analysis (all randomized subjects included), missing data imputed with Expectation Maximization on complete w104 database.
Measure: Count of Participants; unit: Participants
Groups:
- CoBRA Classic High Risk Group: * Methotrexate (MTX)
  * Sulphasalazine
  * Step down steroid full dose
- CoBRA Slim High Risk Group; CoBRA Slim Low Risk Group: * MTX
  * Step down steroid half dose
- CoBRA Avant-garde High Risk Group: * MTX
  * Leflunomide
  * Step down steroid half dose
- Tight Step Up Low Risk Group: * MTX
  * No additional oral steroids allowed
Arm/Group | CoBRA Classic High Risk Group | CoBRA Slim High Risk Group | CoBRA Avant-garde High Risk Group | CoBRA Slim Low Risk Group | Tight Step Up Low Risk Group
Number analyzed (Participants) | 98 | 98 | 93 | 43 | 47
Participants | 69 | 72 | 61 | 25 | 23

2. Primary Outcome: Remission According to DAS28-CRP at Week 52
Description: Number of patients in remission according to DAS28-CRP (Disease Activity Score based on 28 joint count and C-reactive Protein) at week 52. (co-primary end point)
  DAS28-CRP is calculated with the following formula : 0.56*SQRT TJC28+0.28*SQRT SJC28+0.36*ln (CRP+1)+0.014*GH+0.96 in which TJC is the tender joint count, SJC the Swollen Joint Count and GH the general health estimated by the patient on a Visual Analogue Scale (VAS).
  A value below 2.6 is indicating remission, below or equal to 3.2 low disease activity, between 3.2 and 5.1 moderate disease activity and above 5.1 high disease activity.
Time Frame: week 52
Population: ITT (all randomized subjects included), missing data imputed with Expectation Maximization on complete w104 database.
Measure: Count of Participants; unit: Participants
Arm/Group | CoBRA Classic High Risk Group | CoBRA Slim High Risk Group | CoBRA Avant-garde High Risk Group | CoBRA Slim Low Risk Group | Tight Step Up Low Risk Group
Number analyzed (Participants) | 98 | 98 | 93 | 43 | 47
Participants | 63 | 57 | 57 | 29 | 29

3. Primary Outcome: Remission According to DAS28-CRP at Week 104
Description: Number of patients in remission according to DAS28-CRP (Disease Activity Score based on 28 joint count and C-reactive Protein) at week 104. (co-primary endpoints)
  DAS28-CRP is calculated with the following formula : 0.56*SQRT TJC28+0.28*SQRT SJC28+0.36*ln (CRP+1)+0.014*GH+0.96 in which TJC is the tender joint count, SJC the Swollen Joint Count and GH the general health estimated by the patient on a Visual Analogue Scale (VAS).
  A value below 2.6 is indicating remission, below or equal to 3.2 low disease activity, between 3.2 and 5.1 moderate disease activity and above 5.1 high disease activity.
Time Frame: week 104
Population: ITT (all randomized subjects included), missing data imputed with Expectation Maximization on complete w104 database.
Measure: Count of Participants; unit: Participants
Arm/Group | CoBRA Classic High Risk Group | CoBRA Slim High Risk Group | CoBRA Avant-garde High Risk Group | CoBRA Slim Low Risk Group | Tight Step Up Low Risk Group
Number analyzed (Participants) | 98 | 98 | 93 | 43 | 47
Participants | 64 | 71 | 69 | 29 | 34

4. Secondary Outcome: Remission According to SDAI (Simple Disease Activity Index) at Week 16
Description: Number of patients in remission according to SDAI (Simplified Disease Activity Index) at week 16.
  SDAI is calculated with the following formula : TJC28+SJC28+GH+GA ph in which TJC is the number of tender joints, SJC the number of Swollen Joint and GH the general health assessed by the patient on a Visual Analogue Scale (VAS) and GA ph the general assessment of the physician on a VAS.
  A value below 3.3 is indicating remission, between 3.4 and 11.0 low disease activity, between 11.1 and 26.0 moderate disease activity and above 26.0 high disease activity.
Time Frame: week 16
Population: ITT (all randomized subjects included), missing data imputed with Expectation Maximization on complete w104 database.
Measure: Count of Participants; unit: Participants
Arm/Group | CoBRA Classic High Risk Group | CoBRA Slim High Risk Group | CoBRA Avant-garde High Risk Group | CoBRA Slim Low Risk Group | Tight Step Up Low Risk Group
Number analyzed (Participants) | 98 | 98 | 93 | 43 | 47
Participants | 42 | 33 | 44 | 12 | 12

5. Secondary Outcome: Remission According to SDAI at Week 52
Description: Number of patients in remission according to SDAI (Simplified Disease Activity Index) at week 52.
  SDAI is calculated with the following formula : TJC28+SJC28+GH+GA ph in which TJC is the number of tender joints, SJC the number of Swollen Joint and GH the general health assessed by the patient on a Visual Analogue Scale (VAS) and GA ph the general assessment of the physician on a VAS.
  A value below 3.3 is indicating remission, between 3.4 and 11.0 low disease activity, between 11.1 and 26.0 moderate disease activity and above 26.0 high disease activity.
Time Frame: week 52
Population: ITT (all randomized subjects included), missing data imputed with Expectation Maximization on complete w104 database.
Measure: Count of Participants; unit: Participants
Arm/Group | CoBRA Classic High Risk Group | CoBRA Slim High Risk Group | CoBRA Avant-garde High Risk Group | CoBRA Slim Low Risk Group | Tight Step Up Low Risk Group
Number analyzed (Participants) | 98 | 98 | 93 | 43 | 47
Participants | 36 | 27 | 39 | 20 | 15

6. Secondary Outcome: Remission According to SDAI at Week 104
Description: Number of patients in remission according to SDAI (Simplified Disease Activity Index) at week 104.
  SDAI is calculated with the following formula : TJC28+SJC28+GH+GA ph in which TJC is the number of tender joints, SJC the number of Swollen Joint and GH the general health assessed by the patient on a Visual Analogue Scale (VAS) and GA ph the general assessment of the physician on a VAS.
  A value below 3.3 is indicating remission, between 3.4 and 11.0 low disease activity, between 11.1 and 26.0 moderate disease activity and above 26.0 high disease activity.
Time Frame: week 104
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CoBRA Classic High Risk Group | CoBRA Slim High Risk Group | CoBRA Avant-garde High Risk Group | CoBRA Slim Low Risk Group | Tight Step Up Low Risk Group
Number analyzed (Participants) | 98 | 98 | 93 | 43 | 47
Participants | 31 | 28 | 41 | 20 | 13

7. Secondary Outcome: Clinically Significant Change in HAQ Score
Description: Number of patients with a change of > 0.22 in the Health Assessment Questionnaire (HAQ) score over the period between baseline and week 104.
  A change of > 0.22 in this score is considered as clinical relevant for rheumatoid arthritis patients.
Time Frame: Baseline-week104
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CoBRA Classic High Risk Group | CoBRA Slim High Risk Group | CoBRA Avant-garde High Risk Group | CoBRA Slim Low Risk Group | Tight Step Up Low Risk Group
Number analyzed (Participants) | 98 | 98 | 93 | 43 | 47
Participants | 71 | 62 | 64 | 25 | 26

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a two year period per patient
Description: All adverse events were registered by healthcare professionals questioning the patients at each visit
Arm/Group | CoBRA Classic High Risk Group | CoBRA Slim High Risk Group | CoBRA Avant-garde High Risk Group | CoBRA Slim Low Risk Group | Tight Step Up Low Risk Group
All-Cause Mortality (participants affected / at risk) | 1/98 | 1/98 | 0/93 | 0/43 | 0/47
Serious Adverse Events (participants affected / at risk) | 21/98 | 22/98 | 16/93 | 9/43 | 7/47
Other Adverse Events (participants affected / at risk) | 85/98 | 88/98 | 84/93 | 34/43 | 45/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CoBRA Classic High Risk Group (N=98) | CoBRA Slim High Risk Group (N=98) | CoBRA Avant-garde High Risk Group (N=93) | CoBRA Slim Low Risk Group (N=43) | Tight Step Up Low Risk Group (N=47)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone marrow supression (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block third degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus venosus defect (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uncontrolled diabetes mellitus (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Reflux oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylaxis after a wasp sting (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trauma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hernia diaphragmatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Ischialgy leg (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbago (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis flare (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Septic bursitis olecrani (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Baker's cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervixcarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endometrioid adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney cancer malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung cancer malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung noduli (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms parotid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Noduli submandibular salivary glands (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diffuse pain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — induced by MTX
Severe depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peribronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthopaedic surgery (Surgical and medical procedures) | 2 (3) | 1 (1) | 4 (6) | 0 (0) | 1 (1)
Abdominal surgery (Surgical and medical procedures) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Amygdalectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liposuction arms (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolisms (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral vascular ischemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CoBRA Classic High Risk Group (N=98) | CoBRA Slim High Risk Group (N=98) | CoBRA Avant-garde High Risk Group (N=93) | CoBRA Slim Low Risk Group (N=43) | Tight Step Up Low Risk Group (N=47)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 28 (50) | 42 (72) | 29 (46) | 14 (29) | 18 (40)
Abdominal pain (Gastrointestinal disorders) | 25 (27) | 23 (26) | 37 (46) | 11 (14) | 9 (9)
Liver function disturbance (Hepatobiliary disorders) | 17 (22) | 15 (19) | 24 (25) | 6 (6) | 6 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (15) | 7 (8) | 12 (13) | 5 (5) | 3 (4)
Nausea (Gastrointestinal disorders) | 15 (16) | 21 (25) | 12 (14) | 10 (14) | 11 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (13) | 19 (22) | 13 (14) | 3 (4) | 9 (13)
Headache (Nervous system disorders) | 12 (14) | 6 (8) | 9 (12) | 2 (2) | 3 (3)
Vertigo (Nervous system disorders) | 11 (11) | 7 (8) | 6 (7) | 4 (5) | 3 (3)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 10 (10) | 20 (23) | 2 (2) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 13 (14) | 7 (7) | 1 (1) | 1 (1)
General malaise (General disorders) | 9 (9) | 4 (4) | 5 (6) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 9 (9) | 8 (8) | 13 (13) | 4 (4) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 1 (1) | 5 (6) | 2 (2) | 2 (3)
Gastroenteritis (Gastrointestinal disorders) | 8 (9) | 8 (9) | 8 (8) | 8 (9) | 3 (3)
Insomnia (General disorders) | 8 (8) | 4 (4) | 2 (2) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 8 (9) | 3 (3) | 6 (6) | 2 (2) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 7 (8) | 4 (4) | 4 (4) | 2 (2) | 1 (1)
Fatigue (General disorders) | 7 (7) | 4 (6) | 4 (5) | 2 (2) | 5 (5)
Hairloss (General disorders) | 7 (7) | 12 (13) | 19 (20) | 7 (7) | 6 (6)
Increased transpiration (General disorders) | 7 (7) | 3 (3) | 6 (7) | 3 (4) | 1 (1)
Paresthesia (Nervous system disorders) | 7 (9) | 8 (8) | 7 (7) | 3 (3) | 0 (0)
Agitation (General disorders) | 6 (7) | 2 (2) | 10 (10) | 3 (3) | 0 (0)
Flushes (General disorders) | 6 (6) | 4 (4) | 2 (2) | 2 (2) | 0 (0)
Eye infection (Eye disorders) | 6 (8) | 4 (4) | 5 (5) | 1 (1) | 0 (0)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 6 (7) | 5 (6) | 5 (5) | 2 (2) | 4 (4)
Rotator cuff lesion (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Trauma (Injury, poisoning and procedural complications) | 6 (7) | 1 (1) | 6 (7) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 6 (7) | 3 (3) | 7 (9) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 11 (12) | 24 (28) | 1 (1) | 4 (4)
Influenza infection (Infections and infestations) | 5 (6) | 10 (10) | 10 (10) | 2 (3) | 4 (5)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 9 (11) | 12 (12) | 4 (5) | 5 (5)
Tendinopathy (Musculoskeletal and connective tissue disorders) | 5 (5) | 9 (9) | 11 (12) | 5 (5) | 2 (3)
Pyrosis (Gastrointestinal disorders) | 5 (6) | 7 (8) | 2 (2) | 1 (1) | 3 (3)
Aphtosis (Infections and infestations) | 2 (2) | 3 (3) | 8 (10) | 0 (0) | 5 (5)
Genital infection (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 8 (9) | 1 (2) | 0 (0)
Arthrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 6 (6) | 3 (4) | 2 (2)
Sjogren's disease (General disorders) | 5 (5) | 2 (2) | 6 (6) | 2 (2) | 1 (1)
Venous insufficiency (Vascular disorders) | 4 (5) | 5 (5) | 6 (6) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 2 (2)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 4 (4) | 0 (0) | 3 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4) | 5 (5) | 0 (0) | 4 (4)
Renal insufficiency (Renal and urinary disorders) | 1 (1) | 2 (2) | 3 (4) | 0 (0) | 4 (6)
Syncope (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No